CLINICAL TRIAL: NCT01535391
Title: The Protein Tyrosine Kinase Inhibitor Nilotinib as First-line Treatment of Ph+, BCR-, ABL+ Chronic Myeloid Leukemia (CML) in Early Chronic Phase: a Phase IIIb, Multicenter Study to Assess the Complete Molecular Response
Brief Title: Nilotinib in PH+, BCR-, ABL+ CML Patients
Acronym: CML0811
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML0811; 2011-002787-25 (EudraCT Number)
Record Dates: First submitted 2012-02-09; First posted 2012-02-17 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia,; Nilotinib,; Philadelphia positive,; BCR-ABL+; Early chronic phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nilotinib — Administered orally at the dose of 300 mg twice daily (total daily dose 600 mg daily) for 24 months (study core), and indefinitely if it is in the interest of the patient (the drug will be given free-of-charge after 24 months to all those patients achieving the CMR4 at 24 months and in absence of safety concerns). Nilotinib dose is increased to 400 mg BID in case of suboptimal response or failure (with the exception of patients who will fail for progression to ABP: in case of progression to ABP, the patient will not be treated with study drug and the choise of the treatment will be up to the physician).

SUMMARY:
This study is an open-label, multicentric, phase IIIb study of NILOTINIB administered orally twice daily for 24 months and indefinitely if it is in the interest of the patient.

The primary objective of the trial is to evaluate the efficacy of nilotinib, 300 mg twice daily with dose increase to 400 mg twice daily in case of suboptimal response or failure (excluding patients who will fail for progression to ABP), in a population of patients with Ph-positive, BCR-ABL positive CML in early CP.

DETAILED DESCRIPTION:
This study is an open-label, multicentric, phase IIIb study of NILOTINIB administered orally at the dose of 300 mg twice daily (total daily dose 600 mg daily) for 24 months (study core), and indefinitely if it is in the interest of the patient (the drug will be given free-of-charge after 24 months to all those patients achieving the CMR4 at 24 months and in absence of safety concerns). Nilotinib dose is increased to 400 mg BID in case of suboptimal response or failure (with the exception of patients who will fail for progression to ABP: in case of progression to ABP, the patient will not be treated with study drug and the choice of the treatment will be up to the physician).

Study duration is estimated in 6 years, 1 year of estimated enrollment, 2 years therapy duration. Thereafter, information on course and survival is due for other 3 years.

The main data analysis will be performed when all patients will complete 24 months of treatment (or discontinued earlier). Safety and tolerability profile will be assessed by collecting hematologic and non-hematologic adverse events, laboratory examinations and ECG data. The molecular response will be assessed using the GIMEMA standardized molecular laboratories (Labnet network).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Male or female patients with diagnosis of Ph+ and/or BCR-ABL+ CML
* Early chronic phase (within 6 months from diagnosis)
* Pretreatment with Hydroxyurea or Anagrelide for a duration of up to 3 months and/or pretreatment with Imatinib for up to 30 days are permitted
* Normal serum levels of potassium, magnesium, phosphorus, total calcium corrected for serum albumin or phosphorus, or correctable to within normal limits with supplements prior to the first dose of study medication
* Written informed consent prior to any study procedures being performed
* AST and ALT ≤ 2.5 x ULN or ≤ 5.0 x ULN if considered due to leukaemia
* Alkaline phosphatase ≤ 2.5 x ULN unless considered due to leukaemia
* Total direct bilirubin ≤ 1.5 x ULN, except know Mb. Gilbert
* Serum creatinine ≤ 1.5 x ULN

Exclusion Criteria:

* Known impaired cardiac function, including any of the following:
* LVEF < 45%
* Complete left bundle branch block
* Right bundle branch block plus left anterior hemiblock, bifascicular block
* Use of a ventricular-paced pacemaker
* Congenital long QT syndrome
* History of or presence of clinically significant ventricular or atrial tachyarrhythmias
* Clinically significant resting bradycardia (<50 beats per minute)
* QTc>450 msec on screening ECG. If QTc > 450 msec and electrolytes are not within normal ranges before Nilotinib dosing, electrolytes should be corrected and then the patient rescreened for QTc criterion.
* Myocardial infarction within 12 months prior to starting study drugs
* Other clinical significant heart disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension)
* Serum lipase and amylase > 1.5 x ULN (upper limit of normal) or history of acute (i.e., within 1 year of starting study medication) or chronic pancreatitis
* Other concurrent uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infections, acute or chronic liver and renal disease) that could cause unacceptable safety risks or compromise compliance with the protocol
* Impaired gastrointestinal function or disease that may alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting and diarrhea, malabsorption syndrome, small bowel resection or gastric by-pass surgery)
* Concomitant medications with potential QT prolongation (see link for complete list: http://www.torsades.org/medical-pros/drug-lists/printable-drug-list.cfm)
* Concomitant medications known to interact with CYP450 isoenzymes (CYP3A4, CYP2C9,andCYP2C8:link for complete list: http://medicine.iupui.edu/flockhart/table.html..
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are pregnant or breast feeding, or women of reproductive potential not employing an effective method of birth control. (Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to administration of nilotinib).
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Complete molecular response | At 24 months of treatment
  To assess the complete molecular response (CMR4) rate at 24 months of treatment. For the purpose of this protocol, CMR is defined as a negative results of quantitative RT-PCR for BCR-ABL transcripts in a peripheral blood sample of at least 10 ml with a minimum sensitivity of 1:10,000, that corresponds to at least a 4-log reduction (hence, CMR4)

SECONDARY OUTCOMES:
Toxicity | At three years from study entry
  Number of toxic events
Compliance | At 3 years from study entry
  Number of fully compliant patients and number of patients who do not comply with treatment
The complete cytogenetic response (CCgR) rate | At 3, 6, 12, 18 and 24 months from study entry
The rate and the degree of molecular response | At 3, 6, 12, 18 and 24 months from study entry
The time to CCgR, the time to MMR and the time to CMR | baseline
Overall Survival (OS) | At three years from study entry
  From the date of the first nilotinib dose to death
Progression Free Survival (PFS) | At three years from study entry
  From the date of the first nilotinib dose to progression to AP or BP or death
Failure Free Survival (FFS) | At three years from study entry
  From the date of the first nilotinib dose to failure* or progression or death
Event Free Survival (EFS) | At three years from study entry
  From the date of the first nilotinib to any event. Including treatment discontinuation for adverse events, failure, progression to AP or BP, or death, whichever comes first.
Patient-reported quality of life (QoL) | At baseline and then at 3, 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianantonio Rosti, Study Chair — Dpt of Hematology and Oncology, "Seràgnoli", Sant'Orsola-Malpighi. University Hospital of Bologna
Locations (34):
- Italy (34):
  - Azienda Ospedaliera Nuovo Ospedale "Torrette", Ancona
  - S.G. Moscati Hospital, Avellino
  - Azienda Ospedaliera Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - USD Trapianti di midollo per adulti - Cattedra di Ematologia - Università degli Studi di Brescia, Brescia
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Sezione di Ematologia e Fisiopatologia delle Emostasi - Azienda Ospedaliera - Arcispedale S. Anna, Ferrara
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Clinica Ematologica - DiMI - Università degli Studi di Genova, Genova
  - Divisione Ematologia 1 - Azienda Ospedaliera Universitaria "San Martino", Genova
  - U.O. di Ematologia- Ospedale dell'Angelo - Mestre, Mestre
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - Ospedale Cervello, Palermo
  - Azienda Ospedaliera Universitaria - Policlinico Paolo Giaccone, Palermo
  - Div. di Ematologia di Muraglia -CTMO Ospedale San Salvatore, Pesaro
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - IRCCS Centro di riferimento Oncologico di Basilicata, Rionero in Vulture
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Pronto Soccorso e Accettazione Ematologica - Dipartimento Biotecnologie Cellulari ed Ematologia - Università degli Studi di Roma "Sapienza", Roma
  - U.O.C. Ematologia Ospedale S. Eugenio, Roma
  - Università degli Studi Policlinico di Tor Vergata, Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - U.O.C. di Ematolgia - A.O. " SS Annunziata" - P.O. S.G. Moscati, Taranto
  - SCDO Ematologia 2 AOU S.Giovanni Battista, Torino
  - Azienda USL 9 Treviso - U.O. di Ematologia, Treviso
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castagnetti F, Breccia M, Gugliotta G, Martino B, D'Adda M, Stagno F, Carella AM, Avanzini P, Tiribelli M, Trabacchi E, Visani G, Gobbi M, Salvucci M, Levato L, Binotto G, Capalbo SF, Bochicchio MT, Soverini S, Cavo M, Martinelli G, Alimena G, Pane F, Saglio G, Rosti G, Baccarani M; GIMEMA CML Working Party. Nilotinib 300 mg twice daily: an academic single-arm study of newly diagnosed chronic phase chronic myeloid leukemia patients. Haematologica. 2016 Oct;101(10):1200-1207. doi: 10.3324/haematol.2016.144949. Epub 2016 Jul 28. PMID 27470600
- See also: GIMEMA Foundation website — http://www.gimema.it